CLINICAL TRIAL: NCT00635960
Title: Efficacy, Safety and Tolerability of Growth Hormone in Patients With Amyotrophic Lateral Sclerosis as add-on Therapy to Riluzole
Brief Title: Growth Hormone in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Istituto Biostrutture e Immagini, CNR Naples (Unknown); Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Alessandro Filla, Prof., Dipartimento di Scienze Neurologiche, "Federico II" University, Naples
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLA_GH_1
Record Dates: First submitted 2008-03-03; First posted 2008-03-14 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Growth Hormone; IGF-I
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients randomly assigned to treatment
  Interventions: Drug: Growth Hormone (Somatropin)
- 2 (Placebo Comparator): Patients randomly assigned to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Growth Hormone (Somatropin) — The initial dose will be 2U s.c. every other day. The dose will be progressively increased to reach 1.5-2x the normal levels of IGF-I.
  Other Names: Saizen 8mg
  Arms: 1
Drug: Placebo — Same as for Growth hormone group
  Other Names: Saizen 8mg placebo
  Arms: 2

SUMMARY:
Several drugs have been proposed for ALS. These drugs included: Topiramate, Lamotrigine, creatine, Vit. E, Pentoxifylline, etc. Although most of the trials showed a positive trend, none of them reached a statistically significant result. The only exception is the Riluzole trial, that demonstrated a small but significant reduction in mortality between treated and untreated patients. Aim of our study is to determine if the add-on of GH to treatment with Riluzole is able to reduce neuronal loss in the motor cortex of ALS patients.

DETAILED DESCRIPTION:
Several drugs have been proposed for ALS. These drugs included: Topiramate, Lamotrigine, creatine, Vit. E, Pentoxifylline. Although most of the trials showed a positive trend, none of them reached a statistically significant result. The only exception is the Riluzole trial, that demonstrated a small but significant reduction in mortality between treated and untreated patients. When administered to SOD-1 transgenic mice, IGF-I prolongs survival, ameliorates muscular strength, and reduces weight and motor neuron loss, astrocyte gliosis, and ubiquitin positive protein inclusions.

Two clinical trials have been performed in ALS patients with s.c. administration of IGF-I indicating a possible beneficial effect, and a third clinical trial is in progress. Methionyl growth hormone (mGH) showed no effect on survival, disease progression and muscular strength. MGH was administered at a fixed dose and peripheral production of IGF-I appeared to be normal. We propose a double-blind trial of Growth Hormone (GH) as add-on therapy to Riluzole, with an individually regulated dose based on the peripheral response of IGF-I. Aim of our study is to determine if the add-on of GH to treatment with Riluzole is able to reduce neuronal loss in the motor cortex of ALS patients. As secondary objectives, effect of GH on mortality, QoL, and motor function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Definite/probable ALS according to El Escorial criteria
* Aged > 40, < 85 years
* Progression from onset
* Disease duration ≤3 years
* Treatment with Riluzole

Exclusion Criteria:

* Rapid disease progression in the first 6 months after diagnosis
* Patients with tracheostomy and/or Gastrostomy
* Disease duration > 3 years
* Patient with exclusive bulbar or 2° motorneuron involvement
* Hepatic/renal failure
* Pregnant or breastfeeding
* Signs of active neoplasia
* Complicated Diabetes
* Severe hypertension
* Unable to undergo MRI exams

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is the N-acetylaspartate/Creatine ratio in the motor cortex assessed with magnetic resonance spectroscopy. | 0, 6 and 12 months after treatment start

SECONDARY OUTCOMES:
Difference in mortality between groups | 12 months
Difference in the ALS-FRS score (motor function scale) | 0, 6, and 12 months after treatment start
Difference in the SF-36 score (quality of life ) | 0, 6, and 12 monthst after treatmetn start
Safety and tolerability | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Filla, MD, Principal Investigator — University "Federico II", Naples
Locations (2):
- Italy (2):
  - Diparimento di Scienze Neurologiche, Naples
  - Istituto Biostrutture e Bioimmagini, Consiglio Nazionale delle Ricerche, Naples

REFERENCES:
- See also: Institute of Biostructure and Bioimaging, CNR Naples — http://www.ibb.cnr.it/
- See also: University "Federico II", Naples — http://www.unina.it
- See also: Policlinico "Federico II", Naples — http://www.policlinico.unina.it
- See also: AIFA — http://www.agenziafarmaco.it